CLINICAL TRIAL: NCT02977832
Title: A Pilot Study of Clinical Results of Odyliresin (Iresine Celosia) in Symptomatic Benign Prostatic Hyperplasia
Brief Title: Clinical Results of Odyliresin (Iresine Celosia) in Symptomatic Benign Prostatic Hyperplasia
Acronym: Odyliresin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Daniele Porru, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSPSM
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Benign Prostatic Hypertrophy With Outflow Obstruction; Benign Prostatic Hyperplasia
Keywords: LUTS; Iresine celosia; Odyliresin; medical therapy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Intervention Model Description: alpha-antagonist (alfuzosin 10 mg)+ Odyliresin (Iresine celosia) 2 ml, 20 drops once daily.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- odyliresin (Experimental): Odyliresin (Iresine celosia) 2 ml
  Interventions: Dietary Supplement: Odyliresin; Drug: Alfuzosin
- alphalytic (Experimental): alpha-antagonist (alfuzosin 10 mg)
  Interventions: Dietary Supplement: Odyliresin; Drug: Alfuzosin

INTERVENTIONS:
Dietary Supplement: Odyliresin — Odyliresin 2 ml, 20 drops once daily and alpha-antagonist (alfuzosin 10 mg)
  Other Names: Iresine Celosia
Drug: Alfuzosin — 10Mg Oral Tablet, Extended Release
  Other Names: alphalytic

SUMMARY:
Odyliresin (Iresine Celosia) is a cytochrome-flavoprotein with a powerful anti-oxydant action on cells, has a therapeutic effect on BPH-related LUTS, reducing symptoms, prostate volume, improving the patient's quality of life and eventually limiting the number of patients who require surgery or endoscopy after medical treatment.

DETAILED DESCRIPTION:
The aim of this phase II open clinical trial was to determine if Odyliresin, given its unique chemical structure, has a therapeutic effect on BPH-related LUTS, so as to reduce symptoms, prostate volume, improve the patient's quality of life and eventually to limit number of patients who require surgery or endoscopy after medical treatment. To this aim, patients who seek specialist advice for LUTS with no previous surgical treatment for BPH have been selected for treatment with Odyliresin in addition to an alpha-antagonist, in order determine whether at 12 months a clinical result is obtained, if after 6 and 12 months BPH symptoms are significantly improved, and a reduction of prostatic volume can be observed, thus changing the usual course of the disease. All patients with BPH-related LUTS received both alphalitic and Odyliresin treatment, clinical parameters and uroflowmetry parameters significantly improved, adenoma volume and post-void residual volume were significantly reduced at 12 month. This is the first clinical experience with Iresine Celosia in BPH.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or older
* Clinically diagnosed with mild to moderate BPH
* Prostatic volume ≥ 30 ml determined by transrectal ultrasound
* Maximum flow rate (Qmax) < 15 ml/sec for a voided volume 150-500 ml

Exclusion Criteria:

* Participants must not have severe BPH (IPSS symptom score >21)
* Participants should not be currently undergoing any other form of medical therapy for BPH (5-PDE inhibitors, mepartricine, plant extracts such as Saw Palmetto, vitamin E, and quercetin).
* Patients must not have undergone prior transurethral resection of the prostate (TURP).
* Post void residual (PVD) > 200 ml
* Previous urological history including urethral stricture disease and/or bladder neck disease, urinary retention, bladder stone, chronic prostatitis, bladder cancer, interstitial cystitis, active upper tract stone disease causing symptoms, insulin-dependent diabetes mellitus and non-controlled non-insulin-dependent diabetes mellitus, chronic renal failure

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score | 12 months

SECONDARY OUTCOMES:
Maximum flow rate | 12 months
Average flow rate | 12 months
Adenoma volume | 12 months
Residual urine volume | 12 months
adverse events | 12 months
Quality of life score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Tinelli, MD, Study Chair — Ethics Committee
Locations (1):
- Urology Department Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edwards JL. Diagnosis and management of benign prostatic hyperplasia. Am Fam Physician. 2008 May 15;77(10):1403-10. PMID 18533373